CLINICAL TRIAL: NCT01984437
Title: The Robotic Vascular and Endovascular Registry (ROVER)
Brief Title: Registry of the Magellan Robotic System
Acronym: ROVER
Status: Terminated | Type: Observational
Sponsor: Hansen Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: HMP020
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2016-07

CONDITIONS: Peripheral Vascular Disease
Keywords: Vascular disease; Minimally invasive treatment; Endovascular treatment; Magellan; Robotic
MeSH Terms: conditions — Peripheral Vascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the registry is to gather both retrospective and prospective case data on the use of the commercially available Magellan Robotic System and Magellan Robotic Catheters in accordance with the approved intended use. For prospective cases, follow-up patient data will be collected at 14 days (± 5 days) post procedure to assess treatment success, primary patency of intended targeted vessel region, and adverse events.

The data will be analyzed for medical education, societal presentation, and/or publication by the investigators.

Over the next 2+ years, physicians who meet the selection criteria will be invited to participate in the registry.

DETAILED DESCRIPTION:
The objectives of the study are to allow the physician to use the commercially available Magellan Robotic System and Magellan Robotic Catheters to navigate to the treatment targets in the peripheral vasculature to:

* Determine the number of endovascular procedures consecutively performed with the Magellan Robotic System to navigate to treatment targets in the peripheral vasculature and,

  * Achieve stable and efficient system preparation and set-up times, navigation and cannulation times of target vessels during endovascular procedures, and placement of therapeutic equipment used to perform endovascular procedures.
  * Achieve stable and reduced fluoroscopy time during the endovascular procedures.
* Determine the number of cases required to reach a "steady state," reduction or predictable time in conducting peripheral interventional procedures using descriptive (means, ranges) statistics to analyze the data.

Design

This is a prospective and retrospective, multi-center, single arm, non-blinded, sequentially enrolling data collection activity (for which Hansen Medical is providing funding). Only patients scheduled to undergo endovascular procedures using the Magellan Robotic System will be approached for enrollment.

Methods

Registry procedures will be conducted in accordance with the labeled indication for use of the Magellan™ Robotic System.

Prior to the physician participating in the registry and prior to subject enrollment, all participating physicians will be required to complete Hansen Medical's Magellan Robotic System training.

Participating registry sites must have a commercially available Magellan Robotic System for the treatment of patients.

Data Management

Participating sites will be assigned a specific site numeric identification code by the registry sponsor.

The information collected into the registry will be data related to the procedure in which the Magellan System was used or planned to be used and may include patient follow-up data, minimally 14 days(± 5 days)post procedure but also may include 30 day follow-up to assess for the resolution of a procedural or post procedure adverse event.

The database will be a repository for the collected registry data and the data will be made available (in extractable format) to the physician participants.

Adverse Events

The data submitted will be reviewed on a regular basis for safety issues and complaints.

Adverse events and/or complaints deemed reportable will be submitted to the appropriate regulatory agency/agencies by Hansen Medical, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age;
2. Able and willing to provide written informed consent;
3. Eligible for minimally invasive or endovascular treatment in the peripheral vasculature;
4. Not participating in an investigational study involving the peripheral vasculature.

Exclusion Criteria:

1. Disease targeted for treatment in the coronary vasculature or intra-cerebral vasculature;
2. Vasculature that cannot accommodate the Magellan™ Robotic Catheter or required accessories;
3. The required delivery of therapeutic device(s) through the Magellan Robotic Catheter in which the diameter for the therapeutic device(s) is/are incompatible with the Magellan Robotic Catheter;
4. An endovascular approach to the treatment of peripheral vasculature disease is contraindicated.
5. Patients who are prisoners.
6. Patients who are mentally incapacitated, e.g., comatose, unresponsive, cannot provide informed consent, or deemed unreliable or unstable by the investigator.
7. Patients with a cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be diagnosed with vascular disease in the peripheral vasculature, meet all inclusion and no exclusion criteria, and be willing to comply with all protocol testing and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 14 days post procedure
  Consistent manual delivery of therapeutic devices to the target vessel area in the peripheral vasculature by the physician.
Safety | 14 days post procedure
  Incidence and description of device-related (Magellan Robotic System only) adverse events through the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bismuth, MD, Principal Investigator — The Methodist Hospital Research Institute; Brenda Cayme, RN, BSN, Study Director — Hansen Medical, Inc.
Locations (7):
- United States (5):
  - Keck Medical Center of USC, Los Angeles, California
  - Miami Cardiac & Vascular Institute, Miami, Florida
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - The Methodist Hospital, Houston, Texas
- University Hospital of Strasbourg, Strasbourg, France
- Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen, Germany